CLINICAL TRIAL: NCT06490341
Title: Safety and Efficacy of GP Regimen Combined With Nimotuzumab and Sintilimab as Induction Therapy in Locally Advanced Nasopharyngeal Carcinoma: a Single-center, Prospective, Single-arm Phase II Clinical Study
Brief Title: GP Combined With Nimotuzumab and Sintilimab as Induction Therapy for Nasopharyngeal Carcinoma
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NPCTIR001
Record Dates: First submitted 2024-06-29; First posted 2024-07-08 (Actual); Last update posted 2024-07-08 (Actual); Status verified 2024-06

CONDITIONS: Locally Advanced Nasopharyngeal Carcinoma
MeSH Terms: interventions — nimotuzumab; sintilimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- GP Combined with Nimotuzumab and Sintilimab (Experimental): GP regimen(gemcitabine plus cisplatin) in combination with nimotuzumab and sintilimab
  Interventions: Drug: GP Regimen, Nimotuzumab, Sintilimab

INTERVENTIONS:
Drug: GP Regimen, Nimotuzumab, Sintilimab — gemcitabine,ciplatin, nimotuzumab, sintilimab
  Other Names: no other invention names

SUMMARY:
The goal of this clinical trial is to learn if the regimen of gemcitabine, cisplatin combined with nimotuzumab and sintilimab works to treat locally advanced nasopharyngeal carcinoma before chemoradiotherapy. It will also learn about the safety of the regimen. The main questions it aims to answer are:

* Does the regimen increase the number of participants who has a significant tumor shrinkage?
* What medical problems do participants have when taking the regimen? Researchers will evaluate the safety and efficacy of the regimen.

Participants will:

* Take the regimen every 21 days, for twice.
* Visit the clinic weekly for drug administration, checkups and tests.
* Keep a diary of their symptoms.

DETAILED DESCRIPTION:
The study is to investigate the efficacy and safety of combining nimotuzumab and sintilimab with the GP regimen for induction chemotherapy in patients with locally advanced nasopharyngeal carcinoma.

This clinical trial adopts a single-center, prospective, single-arm phase II trial design. Each treatment cycle will be three weeks long, with a total of two cycles.

After screening, eligible patients will be enrolled in the study. Patients will receive two cycles of gemcitabine, cisplatin, nimotuzumab, and sintilimab as induction therapy. Patients will undergo regular follow-up visits, and researchers will collect data on efficacy and safety. Short-term outcomes will be assessed according to the RECIST 1.1 criteria, and adverse events will be evaluated using the CTCAE 5.0.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18 and 75 years, inclusive, without gender restriction.
2. ECOG Performance Status (PS) score of 0 or 1.
3. Histologically confirmed diagnosis of locally advanced nasopharyngeal carcinoma, staged as III-IVa according to the 2018 American Joint Committee on Cancer (AJCC) staging system, with T3-4N2M0 or T1-4N3M0 classification. Tumor types include WHO type II and III.
4. Presence of at least one measurable lesion as per Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1, and patients who have not undergone definitive treatment.
5. Expected survival duration of at least 3 months.
6. White blood cell count ≥ 3 × 10^9/L; absolute neutrophil count ≥ 1.5 × 10^9/L; platelet count ≥ 100 × 10^9/L; hemoglobin level ≥ 90 g/L.
7. Serum creatinine level ≤ 1.2 mmol/L or creatinine clearance ≥ 60 ml/min.
8. Serum total bilirubin ≤ 1.5 × upper limit of normal (ULN) (in case of liver metastasis, ≤ 3.0 × ULN); aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 2.5 × ULN (in case of liver metastasis, ≤ 5.0 × ULN).
9. Female patients must have a negative urine pregnancy test prior to study enrollment (this criterion does not apply to patients with bilateral ovarian resection and/or hysterectomy or postmenopausal patients).
10. Signed written informed consent form.

Exclusion Criteria:

1. Subjects who have received radiotherapy, chemotherapy, immunosuppressive agents, monoclonal antibodies, oral epidermal growth factor receptor tyrosine kinase inhibitors (EGFR-TKIs), or anti-angiogenic drugs within the past six months.
2. Subjects who have participated in another interventional clinical trial, undergone major surgical procedures, or scheduled for surgery within 30 days prior to screening.
3. Patients with severe underlying diseases that preclude tolerance to the treatment.
4. History of other malignancies, except for cured cervical carcinoma in situ, skin basal cell carcinoma, or malignancies cured for more than 5 years without recurrence.
5. Presence of uncontrolled comorbidities such as heart failure, diabetes mellitus, hypertension, thyroid disorders, psychiatric illnesses, etc.
6. Subjects with contraindications to immunotherapy, including those with immune dysfunction diseases (such as rheumatoid arthritis, psoriasis, systemic lupus erythematosus, HIV infection, hepatitis B, hepatitis C, chronic use of steroids for autoimmune diseases), recipients of allogeneic transplants, patients with interstitial lung disease, or those with meningeal metastasis or progressive brain metastasis.
7. Allergy to any of the drugs or their components used in the study protocol.
8. Grade 2 or higher peripheral neuropathy or hearing loss according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) version 5.0.
9. Pregnant women (confirmed by blood or urine human chorionic gonadotropin [HCG] test) or lactating mothers, or subjects of reproductive age who are unwilling or unable to adopt effective contraceptive measures until at least 6 months after the last treatment in the study.

   -

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-07-20 (Estimated); Primary Completion 2026-07-20 (Estimated); Study Completion 2027-07-20 (Estimated)

PRIMARY OUTCOMES:
ORR | 3 months
  objective response rate

SECONDARY OUTCOMES:
mPFS | 1 year
  median progression-free survival
mOS | 2 years
  median overall survival
PFS rate | 3 years
  3-year progression-free survival rate
OS rate | 3 years
  3-year overall survival rate
Adverse events | 1 year
  EGFR and PD-L1 expression, MRD, and others
Radiographic down-staging | 3 months
  stage change according to radiography

CONTACTS AND LOCATIONS:
Overall Officials: He Xiaohui, Principal Investigator — Cancer Hospital, CAMS

IPD SHARING:
Plan to Share IPD: No